CLINICAL TRIAL: NCT03113110
Title: Empagliflozin in Post-Transplantation Diabetes Mellitus
Acronym: EMPTRA-DM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Assoc. Prof. Dr. Manfred Hecking, MD PhD, Assoc. Prof. PD. Dr.med., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EUDRACT-Nr: 2016-001580-37; EK-No. 1366/2016 (Other: MUVienna Ethics Committee)
Record Dates: First submitted 2017-04-08; First posted 2017-04-13 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Posttransplant Diabetes Mellitus
Keywords: Empagliflozin; SGLT-2 Inhibition; Glucose Metabolism
MeSH Terms: interventions — empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Empagliflozin Arm (Other): Posttransplant Diabetes Mellitus (PTDM) patients after kidney transplantation receiving Empagliflozin 10 MG [Jardiance]
  Interventions: Drug: Empagliflozin 10 mg

INTERVENTIONS:
Drug: Empagliflozin 10 mg — PTDM patients on previous antidiabetic treatment (<40 IU insulin (in some cases plus oral antidiabetics)) receive Empagliflozin, ideally as monotherapy
  Other Names: Jardiance

SUMMARY:
RELEVANCE:

Up to 50% of patients without previously known disorders of glucose metabolism develop posttransplantation diabetes mellitus (PTDM) after renal transplantation, which is associated with cardiovascular events. Although PTDM is triggered by immunosuppressive agents (calcineurin inhibitors, glucocorticoids), there is consensus against switching patients from potent tacrolimus to the less diabetogenic cyclosporin. Full-blown PTDM must therefore be treated aggressively. Empagliflozin inhibits sodium-glucose cotransporter 2 in the proximal tubule of the kidney and dramatically reduced cardiovascular risk in type 2 diabetics in a recent randomized trial. Especially in diabetics with impaired renal function, empagliflozin was safe, well tolerated, and effective against hyperglycemia and against high blood pressure. Data on SGLT2 inhibition after transplantation are completely lacking. Therefore, the potential antidiabetic of choice is currently withheld from the vulnerable PTDM population.

METHODS, STUDY DESIGN:

Prospective, single-center, non-inferiority study. Inclusion criteria: PTDM (antidiabetic therapy ≥6 months, based on prior 2-h BG ≥200 mg/dL, fasting BG ≥125 mg/dL (2 times) or HbA1c ≥6.5%); stable renal allograft function >6 months; eGFR ≥30 mL/min/1.73m2. Most important exclusion criteria: type 1 and 2 diabetes; insulin demand >40 IU/day; HbA1c >8.5%. After study inclusion, patients will record 4 weeks of 4-times daily BG measurements before undergoing an OGTT, lab work and urine analysis (including ketones, urinary culture). Empagliflozin (10 mg) will be started and insulin discontinued within 3 days. Patients will be asked to perform urinary dipstick tests at home (i.e. ketones), and to continue recording BG. Study visits at 2 and 4 weeks (second OGTT + lab work (as above)). If control over hyperglycemia is insufficient, insulin therapy will be added back, otherwise study patients remain on empagliflozin monotherapy for 1 year. Statistics will include the paired t-test.

DETAILED DESCRIPTION:
The clinical trial plans to include 16 patients with stable renal allograft function, stable immunosuppressive therapy and PTDM, under standard antidiabetic therapy (exogenous insulin <40 IU). The sample size is based on a calculation assuming non-inferiority of empagliflozin monotherapy in comparison to previous insulin therapy, with respect to the primary endpoint: 2-hour blood glucose (2-h BG) during an oral glucose tolerance test (OGTT) immediately prior and 1 month after the start of empagliflozin monotherapy. The null hypothesis will be accepted if the average change in 2-h BG from the first to the second OGTT exceeds 30 mg/dL (empagliflozin will be inferior). Secondary endpoints comprise the average change in insulin secretory capacity and insulin sensitivity, derived from the first to the second OGTT, the average change in HbA1c at 3 months and at 1 year, compared to baseline, changes in body weight, fluid overload (determined by bioimpedance spectroscopy) and blood pressure. Safety endpoints include clinically concerning hyperglycemia after discontinuation of exogenous insulin, ketoacidosis, urinary tract infections and genital infections, worsening of renal function, hypoglycemia, hospitalizations, cardiovascular events and death. The effect of empagliflozin on the renin-angiotensin system is part of an OeNB-funded project in non-transplanted patients and will be included in the analyses of the present study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed PTDM defined as: A transplant patient requiring antidiabetic therapy, based on a previous 2-hour plasma glucose level ≥ 200 mg/dL in the OGTT (75mg glucose), based on previous blood glucose levels ≥ 200 mg/dL during random controls or based on fasting glucose levels ≥ 125 mg/dL twice or HbA1c ≥ 6.5%
* Stable graft function for more than 6 months post transplantation (eGFR ≥ 30 ml/min/1.73m2)
* At least 6 months of standard of care antidiabetic therapy (usually basal insulin) for PTDM

Exclusion Criteria:

* Age< 18 years
* Patients with prior history of type 1 or type 2 diabetes
* Pregnancy
* Severe renal impairment (GFR < 30 mL/min./1.73 m2)
* Severe blood glucose elevation with the need for therapy with insulin > 40 IU/day or HbA1c >8.5%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2017-01-15 (Actual); Primary Completion 2017-06-13 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
OGTT-derived 2-hour blood glucose level | 4 weeks after start of Empagliflozin treatment
  Mean change from baseline blood glucose levels of the 2h value after OGTT (75g glucose) after 1 month of empagliflozin monotherapy. Maximum tolerable change from baseline blood glucose levels should not exceed 30 mg/dL on average (100 mg/dL in each individual).

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Hecking, MD, Principal Investigator — Department of Internal Medicine III, Division of Nephrology and Dialysis, Medical University of Vienna, Austria
Locations (1):
- Department of Internal Medicine III, Division of Nephrology and Dialysis, Medical University of Vienna, Austria, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schwaiger E, Burghart L, Signorini L, Ristl R, Kopecky C, Tura A, Pacini G, Wrba T, Antlanger M, Schmaldienst S, Werzowa J, Saemann MD, Hecking M. Empagliflozin in posttransplantation diabetes mellitus: A prospective, interventional pilot study on glucose metabolism, fluid volume, and patient safety. Am J Transplant. 2019 Mar;19(3):907-919. doi: 10.1111/ajt.15223. Epub 2019 Jan 25. PMID 30585690